CLINICAL TRIAL: NCT05681689
Title: PyloPlus Urea Breath Test System Post Therapy Efficacy Confirmation Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ARJ Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARJ-2022-UBTPT
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Helicobacter Pylori Infection; Post-Treatment; Efficacy
MeSH Terms: interventions — Shadowing Technique, Histology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Indication for H. pylori testing (Experimental): Patients who have been treated for H. pylori and need to undergo eradication confirmation testing. Patients will be enrolled for this study if all acceptance criteria are met. Patients will undergo 13C Urea Breath Test in addition to non-invasive diagnostic comparators (H. pylori Stool Testing and Comparator Breath Test) OR invasive diagnostic comparator (Endoscopy for Rapid Urease Testing and Histology).
  Interventions: Combination Product: PyloPlus UBT System; Diagnostic Test: Histology; Diagnostic Test: Rapid Urease Test; Combination Product: Comparator Breath Test; Diagnostic Test: Stool Antigen Test

INTERVENTIONS:
Combination Product: PyloPlus UBT System — Breath will be analyzers for change in carbon 13 content in breath after ingestion of enriched carbon 13 urea.
Diagnostic Test: Histology — Biopsy specimen fixed with 10% buffered formalin cut into 4mm sections, stained with Giemsa stain, and examined by experienced pathologist.
Diagnostic Test: Rapid Urease Test — Biopsy specimen obtained and placed onto Rapid Urease Test
Combination Product: Comparator Breath Test — Breath will be analyzers for change in carbon 13 content in breath after ingestion of enriched carbon 13 urea.
Diagnostic Test: Stool Antigen Test — An antigen test performed via a laboratory to test patient's stool for H. pylori

SUMMARY:
This is a multi-center, non-randomized, open label study. Subjects will be enrolled if they are deemed eligible given the inclusion criteria. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. Subjects will be exposed to non-radioactive 13C-Urea with citric acid, and may submit a stool sample or undergo endoscopy for Rapid Urease Test and Histology samples.

Center(s) will house a PyloPlus UBT Analyzer to document results. PyloPlus Analyzer results shall remain blinded to the investigator and treating physician. No patient management decisions should be made based on the investigational PyloPlus UBT System.

Treating physician will either prescribe a H. pylori Stool Antigen Test through P4 Diagnostics, along with another Urea Breath Test using Breath ID, or patient will undergo Endoscopy to provide a composite reference method consisting of Rapid Urease Test and Histology. These will act as the comparators to the PyloPlus Urea Breath Test System.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* Patients who have been diagnosed with H. pylori and have been treated within the past 6 months
* Naive to H. pylori treatment in the past 4 weeks (including PPIs)

Exclusion Criteria:

* Pregnant and/or lactating women.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Participation in other interventional trials.
* Allergy to test substrates.
* Antibiotics taken within 4 weeks of the testing.
* Study subjects shall not consume the following items at least 1 hour prior to the PPUBT test: Mouthwash, Chewing Gum, Carbonated Beverages, Cigarette Smoke, Acetone (to simulate the effect of ketone production that may result from some diets), Alcohol, Food

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Overall Percent Agreement | 7 days
  The primary study endpoint is the performance measure on H. pylori eradication confirmation via PyloPlus Urea Breath Test and Comparators

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dolphin Medical Research, Doral, Florida
  - Hudson County Clinical Trials Research Center, Union City, New Jersey

IPD SHARING:
Plan to Share IPD: No